CLINICAL TRIAL: NCT04718584
Title: A Single-arm, Open, Multicenter, Phase II Clinical Study of the Efficacy and Safety of Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) in the Treatment of Urinary and Male Genital Tumors
Brief Title: the Efficacy and Safety of LDP in Patients With Urinary and Male Genital Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDP-II-01
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Bladder Cancer; Renal Carcinoma; Advanced Penile Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arms (Experimental): All participants will receive treatment with LDP 10mg/kg once every two weeks, every 2 weeks will be a cycle. In Cort 1, surgical treatment will be performed within 2 weeks after the end of 3 cycles of treatment.
  Interventions: Drug: Human Anti-PD-L1 Monoclonal Antibody Injection (LDP)

INTERVENTIONS:
Drug: Human Anti-PD-L1 Monoclonal Antibody Injection (LDP) — All participants will receive treatment with LDP 10mg/kg once every two weeks, every 2 weeks will be a cycle. In Cort 1, surgical treatment will be performed within 2 weeks after the end of 3 cycles of treatment.
  Other Names: LDP

SUMMARY:
This is a single-arm,open, multicenter, phase II clinical study of the efficacy and safety of human anti-PD-L1 monoclonal antibody Injection (LDP) in the treatment of urinary and male genital tumors.

DETAILED DESCRIPTION:
This trial is a single arm, open, multicenter, Ⅱ period clinical research. Three cohorts were included, 127 subjects were enrolled (Cohort 1: about 60 subjects with surgically suitable muscular-invasive bladder cancer; Cohort 2: about 40 subjects with advanced Non-clear Cell Renal Carcinoma; Cohort 3: about 27 subjects with advanced penile carcinoma. After confirmation of inclusion, intravenous infusion of 10mg/kg human anti-PD-L1 monoclonal antibody injection (LDP) was given. The initial efficacy and safety of drugs in different tumor species in the cohort above will be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 (inclusive), ≤18 (inclusive)
2. Patients with muscular-infiltrating bladder cancer suitable for surgery; advanced opaque cell renal carcinoma; advanced penile carcinoma
3. The estimated survival time is more than 3 months.
4. At least one assessable tumor lesion according to RECIST1.1 (in cohort 1, evaluate lesion is accept);
5. ECOG physical strength score 0-1;
6. Enough organ function: Blood routine (no blood transfusion or colony stimulating factor (G-CSF) treatment within 14 days):ANC≥1.5×109 / L, PLT≥75×109 / L, Hb≥80g/L; Liver function: TBIL≤1.5×ULN, ALT≤2.5×ULN, AST≤2.5×ULN (ALT,AST≤5×ULN for liver metastasis patients); Renal function: Cr ≤ 1.5 × ULN, and creatinine clearance > 50 ml /min(according to Croft Gault formula) ; Coagulation function: APTT≤ 1.5 ×ULN, PT ≤ 1.5 × ULN, INR ≤ 1.5 × ULN;
7. Eligible patients (male and female) with fertility must agree to use reliable methods of contraception (hormone or barrier or abstinence) during the trial period and at least 6 months after the last dose; The blood or urine pregnancy test within 7 day before being selected must be negative for the female patients of childbearing age;
8. Subjects must give informed consent to this study before the study, and voluntarily sign a written informed consent;

Exclusion Criteria:

1. Received radiotherapy, chemotherapy, targeted therapy, endocrine therapy or immunotherapy within 4 weeks before the first administration, or other unlisted clinical trial drug therapy (mitomycin and nitrosourea are 6 weeks from the last administration, oral fluorouracil drugs such as Tegiol and Capecitabine are at least 2 weeks from the last administration, small molecule targeted drugs are at least 2 weeks or at least interval 5 half-life (Subject to the longer time) from the last administration, and traditional Chinese medicine with antitumor indications are at least 2 weeks from the last administration.
2. Major organ surgery (excluding puncture biopsy) or significant trauma occurred within 4 weeks prior to the first administration.
3. The adverse effects of previous antitumor therapy have not recovered to CTCAE 5.0 ≤grade1 (except for alopecia)
4. Patients with clinical symptoms of brain metastases, spinal cord compression, cancerous meningitis, or other evidence of uncontrolled brain or spinal cord metastases are not suitable for inclusion as judged by the investigator
5. Patients who had previously received PD-1 or PD-L1 inhibitors;
6. Immunorelated adverse events ≥ Grade 3 were observed in previous immunotherapy except for PD-1 or PD-L1 inhibitors;
7. Patients have any active autoimmune diseases or a history of autoimmune diseases (e.g., but not limited to: systemic lupus erythematosus, autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, vitiligo, etc.); Complete remission of asthma in childhood can be included if in adults without any intervention;Asthma patients requiring bronchodilators for medical intervention were excluded);
8. Patients who received systemic corticosteroid (prednisone > 10mg/ day or equivalent) or other immunosuppressive therapy within 14 days prior to initial dosing; Exceptions include: topical, ocular, intraarticular, intranasal, and inhaled corticosteroids;Short-term use of corticosteroids for preventive treatment, such as before the use of contrast agents;
9. Malignancies that were active within the last 2 years prior to initial administration (except for the tumors targeted in this study);
10. Uncontrolled active hepatitis B (HBsAg positive with HBV DNA copy number > 103/ mL or HBV DNA titer >200 IU/ mL); Hepatitis C;
11. Syphilis infection (syphilis antibody positive) and HIV positive patients.
12. A history of serious cardiovascular disease, including ventricular arrhythmias requiring clinical intervention;Acute coronary syndrome, congestive heart failure, stroke, or other grade 3 or higher cardiovascular events within 6 months;New York Heart Association (NYHA) cardiac function grade ≥II or left ventricular ejection fraction (LVEF) < 50%;Patients with clinically uncontrolled hypertension who are not suitable for the trial as determined by the investigator;
13. Patients with a history of other serious systemic diseases who have been determined by the investigator to be unsuitable for participation in clinical trials;
14. Known alcohol or drug dependence;
15. Mental disorder or poor compliance;
16. Women who are pregnant or lactating;
17. Have received live attenuated vaccine within 4 weeks before the first administration or scheduled to receive during the study period.
18. The Investigator considers that the subject is unsuitable to participate in this study because of any clinical or laboratory test abnormalities or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Case complete response （pCR） | At the end of the cycle 3 of treatment (each cycle is 14 days).
  The pCR is defined as the case complete response in Cohort 1 (muscular-infiltrating bladder cancer suitable for surgery)
Objective response rate (ORR) | From first dose of LDP through 21 days after last dose of LDP up to 2 years.
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1 in Cohort 2 (Non-clear Cell Renal cell Carcinoma) and Cohort 3 (advanced penile carcinoma)

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | One year after surgery or disease progression or intolerant toxicity, up to 2 years.
  Recurrence-free survival (RFS) is defined as the time from the start of surgery to the earliest evidence of recurrence.
Progression-free survival （PFS） | From first dose of LDP, up to 2 years.
  Progression-free survival (PFS) is defined as the time elapsed from the day the study drug was first administered until the first imaging assessment of disease progression (PD) or death from any cause.
Disease control rate (DCR) | From first dose of LDP, up to 2 years.
  Disease control rate (DCR) is defined as the proportion of the optimal time response of CR, PR, disease stable (SD) (i.e. CR+PR+SD) between initiation of the trial drug and withdrawal from the trial, as assessed according to RECIST1.1 criteria.
Duration of response (DOR) | From first dose of LDP, up to 2 years.
  The duration of response (DOR) is defined as the time from the beginning of the first tumor assessment as PR or CR to the first assessment as PD or death from any cause.
Overall survival (OS) | From first dose of LDP, up to 2 years.
  Overall survival (OS) is defined as the time between the date of first use of the study drug and death from any cause.
Incidence of adverse events | From first dose of LDP through 30 days after last dose of LDP, up to 5 months.
  Adverse events (AEs) refer to all adverse medical events that occur when subjects sign the informed consent, which may be manifested as symptoms, signs, diseases or abnormal laboratory tests, but not necessarily causally related to the investigational drug.
Incidence of abnormal vital signs | From first dose of LDP through 30 days after last dose of LDP, up to 5 months.
  Vital signs (including temperature, respiration, heart rate and blood pressure) can be measured. The time window for each vital sign measurement is ±10 minutes.
Incidence of abnormal ECOG scores | From first dose of LDP through 30 days after last dose of LDP, up to 5 months.
  ECOG physical strength rating is based on ECOG physical strength rating criteria.
Incidence of abnormal laboratory tests results | From first dose of LDP through 30 days after last dose of LDP, up to 5 months.
  Descriptive analysis of laboratory results for safety analysis.
Incidence of abnormal physical examinations | From first dose of LDP through 30 days after last dose of LDP, up to 5 months.
  Descriptive analysis of physical examination for safety analysis.
anti-drug antibody (ADA) | In Cohort 1: before administration ,before surgery; In Cohort 2, 3: before administration, up to 4 months.
  Anti-drug antibody (ADA) is tested for immunogenicity assessment , titer and neutralizing antibody analysis were performed when ADA was positive, and immunocomplex (CIC) and complement analysis were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Study Chair — Fudan University
Locations (1):
- Dragonboat Biopharmaceutical,Co.,Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No